CLINICAL TRIAL: NCT04476407
Title: "Pharmacokinetics of Benapenem in Subjects With Mild or Moderate Renal Impairment "
Brief Title: Pharmacokinetics of Benapenem in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5081-I-1004
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2019-04

CONDITIONS: Complicated Urinary Tract Infection; Cuti
MeSH Terms: interventions — benapenem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1 (Experimental): subjects with nomal renal function
  Interventions: Drug: benapenem
- G2 (Experimental): subjects with mild renal impairment
  Interventions: Drug: benapenem
- G3 (Experimental): subjects with moderate renal impairment
  Interventions: Drug: benapenem

INTERVENTIONS:
Drug: benapenem — single-dose Benapenem 1.0mg(iv), 60min infusion
  Arms: G1
Drug: benapenem — single-dose Benapenem 1.0mg(iv), 60min infusion
  Arms: G2
Drug: benapenem — single-dose Benapenem 1.0mg(iv), 60min infusion
  Arms: G3

SUMMARY:
This is an open-label, multiple center, parallel-group Study to compare the pharmacokinetics and safety of single-dose benapenem (1.0mg) in subjects with mild or moderate Renal Impairment(RI) and healthy subjects. Subjects were enrolled with defined degrees of RI based on eGFR(estimated Glomerular Filtration Rate) calculated by MDRD (Modification of Diet in Renal Disease)formular as follows: nomal renal function(≥90ml/min/1.73m2 ; N=6); mild RI (60-89mL/min/1.73 m2 ; N=6), moderate RI (30-59 mL/min/1.73m2 ; N=6)

ELIGIBILITY:
Inclusion Criteria:

* 1.18~75 years old
* 2. BMI 17 to 30 kg/m2
* 3. No known diseases or significant abnormalities on physical exam (subjects with normal renal function only)
* 4. eGFR ≥ 90 mL/min/1.73m2 (subjects with normal renal function only)
* 5. eGFR 30 to 59 mL/min/1.73m2 (subjects with mild renal impairment only); eGFR 60 to 89 mL/min/1.73m2 (subjects with moderate renal impairment only)

Exclusion Criteria:

* 1. Hypersensitivity to any of the beta-lactam antibiotics
* 2.Conditions or disease that may interfere with the evaluation of study drug
* 3. Acute disease requiring antibiotics within 30 days prior to administration, or a fever within 7 days prior to administration;
* 4. Drug abuse in 2 years
* 5. A blood donation or more than 400 ml of blood loss within 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | predose and 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 hours postdose
  Area under the plasma concentration-time curve from time 0 to the time of thelast quantifiable concentration (AUC0-t )of benapenem and the metabolite
Area under the plasma concentration-time curve | predose and 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 hours postdose
  Area under the plasma concentration-time curve from time 0 to infinity ( AUC0-inf ) of benapenem and the metabolite
Maximum observed plasma concentration(Cmax) | predose and 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48, 72 hours postdose
  Maximum observed plasma concentration(Cmax) of benapenem and the metabolite
Observed terminal elimination half-life (T1/2) | predose, 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48 and 72 hours postdose
  Observed terminal elimination half-life (T1/2) of benapenem and its metabolite
Total body clearance (CLt) | predose, 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48 and 72 hours postdose
  Total body clearance (CLt) of benapenem
Apparent volume of distribution (Vz) | predose, 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48 and 72 hours postdose
  Apparent volume of distribution (Vz) based on the terminal phase of benapenem
Cumulative urine exeretion | predose, 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48 and 72 hours postdose
  Cumulative urine exeretion (Ae0-72h%) of benapenem and its metabolite
Renal clearance (CLr) | predose, 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48 and 72 hours postdose
  Renal clearance (CLr) of Benapenem and its metabolite
Metabolite-to-parent ratio of AUC0-inf | predose, 0.5, 1.25, 1.5, 2, 3, 5, 8, 12, 24, 48 and 72 hours postdose
  Metabolite-to-parent ratio of AUC0-inf (MR)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China